CLINICAL TRIAL: NCT03204994
Title: Investigating the Feasibility of Fluorescence Targeted Pelvic Lymph Node Mapping During Rectal Cancer Surgery
Brief Title: Fluorescence Targeted Pelvic Lymph Node Mapping
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Not able to recruit
Sponsor: Oxford University Hospitals NHS Trust (Other)
Responsible Party: Principal Investigator, Thomas Barnes, Clinical Research Fellow, Oxford University Hospitals NHS Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12451
Record Dates: First submitted 2017-06-28; First posted 2017-07-02 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Cancer of Rectum; Lymph Node Disease
Keywords: Colorectal surgery; Fluorescence guided surgery
MeSH Terms: conditions — Rectal Neoplasms | interventions — Indocyanine Green

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tumour injection of ICG (Experimental): Indocyanine green injection into tumour before or during surgery.
  Interventions: Drug: Indocyanine Green

INTERVENTIONS:
Drug: Indocyanine Green — Fluorescence guided lymphatic mapping using indocyanine green.
  Other Names: ICG

SUMMARY:
This study aims to assess the lymphatic drainage of rectal tumours by using ICG as a fluorescent non-specific marker. As a feasibility study, it will also assess its technique and timing along with its ability to assist in removing lymph nodes when it is clinically indicated.

DETAILED DESCRIPTION:
Current surgical treatment for rectal cancer includes total mesorectal excision (TME) which involves excision of the rectum in its encompassing fat including the lymph nodes. Rectal cancer can spread to lymph nodes locally inside the TME 'package' and the lateral pelvic lymph nodes. The TME must be fully excised to ensure that the circumferential resection margin (CRM) is disease free or negative. Despite advancing surgical techniques, a positive margin can occur in around 9% of patients with accurate pre-operative magnetic resonance imaging (MRI), increasing the risk of local recurrence.

Incidence of lateral pelvic lymph node involvement has been reported between 10-25%. It is thought that lower rectal tumours are more likely to spread to the lateral pelvic nodes. In the far East, LPLN dissection is often added to the TME procedure. Formal LPLND is not utilised in Europe due to operative risks including damage to pelvic nerves, greater blood loss and prolonged operating time. Instead, neoadjuvant chemoradiotherapy (CRT) is utilised to 'sterilise' the lymph nodes. Although a retrospective analysis suggested that LPLN dissection is equivalent to preoperative CRT for preventing local recurrence, there has been evidence to suggest that positive LPLNs after CRT decrease cancer specific survival and relapse free survival. This would suggest that there may be a cohort of patients that would benefit from some form of LPLN dissection, although it is not certain what characteristics of tumours are more likely to metastasise to the LPLNs.

In prostatectomies, where pelvic lymph node dissection is a standard part of the procedure, there has been investigation into fluorescence guided lymph node mapping. Yuen et al utilised ICG guided node mapping in open prostatectomy. In their study, all lymph nodes identified by fluorescence were found to have metastases on pathology whereas non-fluorescent nodes were free from disease. A smaller, retrospective study comparing fluorescence guided lymph node dissection with standard lymph node dissection showed higher sensitivity and specificity in the fluorescence guided technique. Similar results were seen in an early, robotic prostatectomy study.

ICG has been used to map pelvic lymph nodes in colorectal cancer, with the first reported cases being published in 2010. ICG was injected to the tumour base in 25 open rectal resections. A wide field camera is useful for fluorescence in open surgery, however, as most rectal cancer cases are performed using a minimally invasive approach a laparoscopic method is needed. Ishizuka et al used a similar method in low rectal cancers to identify drainage in three different sets of lymph nodes. In 2015, a study of 5 patients using ICG node mapping with the same laparoscopic equipment to be used in this study demonstrated fluorescence in all 5 patients. Both studies 'berry picked' the fluorescing lymph nodes. In the 2010 study, 23 out of 25 patients had fluorescing lymph nodes. In the 2 non-fluorescing nodes LPLD was performed and no diseased nodes were identified. In these studies, they did not observe what types of tumours drain to the LPLDs.

ICG, when injected intravenously, rapidly binds to plasma proteins and is exclusively excreted into bile by the liver. It is known to be well tolerated but there have been reported cases of urticaria and anaphylaxis. Risk of anaphylaxis is 1 in 10,000 and if occurs can be treated using a standard protocol. ICG contains sodium iodide and therefore should be avoided in patients with known allergy to iodides.

This study aims to assess the lymphatic drainage of rectal tumours by using ICG as a fluorescent non-specific marker. As a feasibility study, it will also assess its technique and timing along with its ability to assist in removing lymph nodes when it is clinically indicated.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Male or Female, aged 18 years or above.
* Participant is undergoing elective curative surgery for rectal adenocarcinoma
* Participant is willing and able to comply with study requirements

Exclusion Criteria:

* Participant has history of or known allergy to indocyanine green
* Participant has history of or known allergy to iodides
* Participant suffers from hyperthyroidism or has a benign thyroid tumour
* Participant has renal failure
* Female participant currently pregnant, planning pregnancy or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Number & location of lymph nodes identified with and without fluorescent probe during rectal cancer surgery | 1 day

SECONDARY OUTCOMES:
Noise to background signal of lymph nodes compared with positivity of lymph nodes. | 1 day
  Positivity defined as whether they contain metastatic disease or not.
Number of lymph nodes lying outside the CRM identified by fluorescence | 1 day
  Fluorescence identification of CRM nodes

CONTACTS AND LOCATIONS:
Overall Officials: Chris Cunningham, MD, Principal Investigator — Chief Investigator; Thomas Barnes, MBChB, Principal Investigator — Clinical Research Fellow
Locations (1):
- Oxford University Hospitals NHS Foundation Trust, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No